CLINICAL TRIAL: NCT02261090
Title: A Multiple Dose Seven-way Cross-over Formulation-finding Study Comparing the Oral Bioavailability of Seven Prototype Slow-release Formulations With 0.75 mg Pramipexole (Four Days Each) to Immediate-release Tablets at Steady State in Healthy Male Volunteers
Brief Title: Bioavailability of Different Pramipexole Slow-release Formulations Compared to Immediate-release Tablet in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 248.529
Record Dates: First submitted 2014-10-09; First posted 2014-10-10 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Tablets; Pramipexole

ARMS (8):
- Formulation B (Experimental): Slow release (SR) tablet
  Interventions: Drug: Formulation B: Pramipexole Slow release (SR) tablet
- Formulation C (Experimental): SR tablet
  Interventions: Drug: Formulation C: Pramipexole Slow release tablet
- Formulation D (Experimental): SR tablet
  Interventions: Drug: Formulation D: Pramipexole Slow release tablet
- Formulation E (Experimental): SR tablet
  Interventions: Drug: Formulation E: Pramipexole Slow release tablet
- Formulation F (Experimental): SR tablet
  Interventions: Drug: Formulation F: Pramipexole Slow release tablet
- Formulation G (Experimental): SR tablet
  Interventions: Drug: Formulation G: Pramipexole Slow release tablet
- Formulation H (Experimental): SR tablet
  Interventions: Drug: Formulation H: Pramipexole Slow release tablet
- immediate release (IR) formulation (Active Comparator)
  Interventions: Drug: Pramipexole immediate release (IR) tablets

INTERVENTIONS:
Drug: Formulation B: Pramipexole Slow release (SR) tablet
  Arms: Formulation B
Drug: Formulation C: Pramipexole Slow release tablet
  Arms: Formulation C
Drug: Formulation D: Pramipexole Slow release tablet
  Arms: Formulation D
Drug: Formulation E: Pramipexole Slow release tablet
  Arms: Formulation E
Drug: Formulation F: Pramipexole Slow release tablet
  Arms: Formulation F
Drug: Formulation G: Pramipexole Slow release tablet
  Arms: Formulation G
Drug: Formulation H: Pramipexole Slow release tablet
  Arms: Formulation H
Drug: Pramipexole immediate release (IR) tablets
  Arms: immediate release (IR) formulation

SUMMARY:
Study to compare the oral bioavailability of seven prototype slow-release formulations to immediate-release tablets

ELIGIBILITY:
Inclusion Criteria:

* All participants in the study should be healthy males
* Participants should be ranging from 21 to 50 years of age
* Body mass index (BMI) within 18.5 to 29.9 kg/m2
* In accordance with Good Clinical Practice and the local legislation all volunteers will have given their written informed consent prior to admission to the study

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24:00 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study or during the study
* Use of any drugs which might influence the results of the trial up to 7 days prior to enrolment in the study or during the study
* Participation in another trial with an investigational drug (≤ two months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on in-house trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (≥ 100 mL within four weeks prior to administration or during the trial)
* Any laboratory value outside the clinically accepted reference range
* Excessive physical activities within the last week before the trial or during the trial
* Hypersensitivity to pramipexole, or other dopamine agonists
* Supine blood pressure at screening of systolic < 110 mmHg and diastolic < 60 mmHg
* A haemoglobin value at screening of less than 13.5 g/dl (usual lower limit of normal for males: 12.6 g/mL)
* Subjects involved in passenger transport or operation of dangerous machines

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2004-06; Primary Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Plasma total exposure (AUCτ,ss) | up to 168 hours after each drug administration
Urine total exposure (Aeτ,ss) | up to 168 hours after each drug administration
Plasma maximum exposure (Cmax,ss) | up to 168 hours after each drug administration
Plasma minimum exposure (Cmin,ss) | up to 168 hours after each drug administration
Plasma average concentration (Cavg) | up to 168 hours after each drug administration
Plasma peak to trough fluctuation (PTF) | up to 168 hours after each drug administration

SECONDARY OUTCOMES:
AUC0-6,11 for the immediate release (IR) formulation | day 7 of visit 2
Cmax for the IR formulation | up to 168 hours after drug administration in visit 2
Cmin for the IR formulation | up to 168 hours after drug administration in visit 2
tmax for the IR formulation | up to 168 hours after drug administration in visit 2
Urinary excretion (Ae) for the IR formulation | up to 168 hours after drug administration in visit 2
tmax,4 for the SR formulation | up to 96 hours after drug administration in visit 3-5, 7 and 9
t1/2,4 for the SR formulation | up to 96 hours after drug administration in visit 9
Urinary excretion (Ae) for the SR formulation | up to 168 hours after drug administration
Number of subjects with adverse events | up to 8 days after last drug administration
Number of subjects with clinically significant findings in laboratory tests | up to 8 days after last drug administration
Number of subjects with clinically significant findings in vital signs | up to 8 days after last drug administration
  blood pressure, pulse rate
Assessment of global tolerability by investigator on a 5-point scale | at the end of each of the visits 2 to 9